CLINICAL TRIAL: NCT01039948
Title: A Phase 1b/2 Study of AV-299 (Formerly SCH 900105) in Combination With Gefitinib in Asian Subjects With Non-Small Cell Lung Cancer (P06162)
Brief Title: A Phase 1b/2 Study in Asian Subjects With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AVEO Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P06162
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Carcinoma, Non-Small Cell-Lung; Lung Neoplasms; Lung Cancer; Respiratory Tract Neoplasms
Keywords: Neoplasms; Carcinoma; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Respiratory Tract Neoplasms; Neoplasms, Glandular and Epithelial; Neoplasms by Histological Type; Thoracic Neoplasms; Neoplasms by Site; Lung Diseases; Respiratory Tract Diseases; Gefitinib; Antineoplastic Agents; Therapeutic Uses; Pharmacologic Actions; Protein Kinase Inhibitors; Enzyme Inhibitors; Molecular Mechanisms of Pharmacological Action
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Respiratory Tract Neoplasms; Neoplasms; Carcinoma; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Thoracic Neoplasms; Neoplasms by Site; Lung Diseases; Respiratory Tract Diseases | interventions — ficlatuzumab; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase 2: AV-299 + gefitinib (Experimental): Phase 2: AV-299 (formerly SCH 900105) administered IV at RP2D (as determined by Phase 1b portion) in combination with gefitinib 250 mg/day orally.
  Interventions: Biological: AV-299 + gefitinib
- Phase 2: Gefitinib (Active Comparator): Phase 2: Gefitinib 250 mg/day, orally.
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Biological: AV-299 + gefitinib — AV-299 is a humanized anti-HGF IgG1 monoclonal antibody directed against free HGF, ligand for c-Met tyrosine kinase receptor.
  Other Names: Other name: ficlatuzumab, Formerly SCH 900105
  Arms: Phase 2: AV-299 + gefitinib
Drug: Gefitinib — Gefitinib is a small molecule (drug) which selectively inhibits epidermal growth factor receptor's (EGFR) tyrosine kinase domain.
  Other Names: Iressa®
  Arms: Phase 2: Gefitinib

SUMMARY:
During Phase 1b portion, there will be a dose-escalation of AV-299 (formerly SCH 900105) in combination with the recommended dose of gefitinib in subjects with NSCLC or advanced solid tumor. The objective is to determine the safety, tolerability, dose limiting toxicity (DLT) and recommended Phase 2 dose (RP2D) in combination with gefitinib for the Phase 2 portion.

The Phase 2 is an open-label, 2-arm, randomized study designed to compare the combination of AV-299 (formerly SCH900105) and gefitinib versus gefitinib alone in clinically selected Asian subjects with previously untreated lung adenocarcinoma who have a high likelihood of harboring activating EGFR mutations. Subjects who progress after initial disease control in the gefitinib alone arm may crossover to the combination arm.

ELIGIBILITY:
Inclusion Criteria:

* Asian ethnicity.
* ECOG performance status of 0-2.
* Phase 1b (only): Diagnosis of one of the following unresectable NSCLC with or without prior therapy advanced solid tumor that progressed after standard therapy
* Phase 2 only: Histologic or cytologic confirmation of unresectable locally advanced or metastatic stage IIIB/IV lung adenocarcinoma with at least one measurable lesion, per Response Evaluation Criteria in Solid Tumors (RECIST-Version 1.1).
* Phase 2 only: Never smoker or light ex-smoker.
* Available tumor tissue for determination of EGFR mutational status and immunohistochemistry analysis
* Adequate hematologic, hepatic, renal and coagulation function
* No active central nervous system metastases
* Prior radiotherapy is allowed if 14 days from first dose of study drug and toxicity is resolved; additionally in Phase 2 only, ≥1 target lesion not irradiated or with definitive progression after prior radiation therapy.
* Agreement to use effective contraception.
* Phase 2 only: Subjects on Gefitinib monotherapy arm must have documented CR, PR, or SD for ≥12 weeks prior to disease progression in order to cross over to combination therapy arm.

Exclusion Criteria:

* Phase 2 only: Prior chemotherapy or prior treatment with epidermal growth factor receptor (EGFR) inhibitor, including both tyrosine kinase inhibitors and monoclonal antibodies. There is no limit to the number of therapies for subject being considered for Phase 1b.
* History of neoplasm other than the entry diagnosis.
* Pregnancy or lactation.
* Myocardial infarction within 6 months prior to initiation of study treatment.
* A serious active infection.
* Known human immunodeficiency virus infection.
* A serious underlying medical condition that would impair the ability of the subject to receive protocol treatment.
* A major surgical procedure, open biopsy, or significant traumatic injury.
* Thrombotic or embolic events.
* Known or suspected allergy/hypersensitivity to any agent given in the course of this trial.
* Any condition that impairs absorption of oral agents or the subject's ability to swallow whole pills.
* Diarrhea ≥ Grade 2 or active Inflammatory Bowel Disease.
* Severe acute or chronic medical, psychiatric, or behavioral condition or laboratory abnormality.
* Diagnosis of interstitial lung disease.
* Any medications or treatments prohibited by the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2009-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Phase Ib: Dose Limiting Toxicity and Recommended Phase II Dose | Every 4 weeks for the first 4 months of treatment period, every 8 weeks thereaftert
Phase 2: Objective Response Rate | Every 4 weeks for the first 4 months of treatment period, every 8 weeks thereafter

SECONDARY OUTCOMES:
Phase 1b: Cmax, Tmax, AUC, t1/2, clearance, and Vd | Every 4 weeks for the first 4 months of treatment period, every 8 weeks thereafter
Phase 2: Progression Free Survival, Overall Survival, Safety | Every 4 weeks for the first 4 months of treatment period, every 8 weeks thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Philip Komarnitsky, MD, Study Director — AVEO Pharmaceuticals, Inc.
Locations (26):
- Investigational Site 1, Shatin N.T., Hong Kong
- Malaysia (3):
  - Investigational Site 10, Kuala Lumpur
  - Investigational Site 9, Kuala Lumpur
  - Investigational Site 11, Kuala Pahang
- Philippines (3):
  - Investigational Site 12, Manila
  - Investigational Site 13, Pasig
  - Investigational Site 14, Quezon City
- Investigational Site 15, Singapore, Singapore
- South Korea (7):
  - Investigational Site 2, Chungcheongbuk-do
  - Investigational Site 3, Gyeonggi-do
  - Investigational Site 4, Jeollanam-do
  - Investigational Site 5, Seoul
  - Investigational Site 6, Seoul
  - Investigational Site 7, Seoul
  - Investigational Site 8, Seoul
- Taiwan (7):
  - Investigational Site 16, Changhua
  - Investigational Site 17, Chiayi City
  - Investigational Site 18, Taichung
  - Investigational Site 19, Tainan
  - Investigational Site 20, Taipei
  - Investigational Site 21, Taipei
  - Investigational Site 22, Taoyuan District
- Thailand (4):
  - Investigational Site 23, Bangkok
  - Investigational Site 24, Chiang Mai
  - Investigational Site 25, KhonKaen
  - Investigational Site 26, Songkhla

REFERENCES:
- [Derived] Tan EH, Lim WT, Ahn MJ, Ng QS, Ahn JS, Shao-Weng Tan D, Sun JM, Han M, Payumo FC, McKee K, Yin W, Credi M, Agarwal S, Jac J, Park K. Phase 1b Trial of Ficlatuzumab, a Humanized Hepatocyte Growth Factor Inhibitory Monoclonal Antibody, in Combination With Gefitinib in Asian Patients With NSCLC. Clin Pharmacol Drug Dev. 2018 Jun;7(5):532-542. doi: 10.1002/cpdd.427. Epub 2018 Jan 18. PMID 29346833